CLINICAL TRIAL: NCT00611936
Title: Effects of Atomoxetine Treatment in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0605001441
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Stress
Keywords: Atomoxetine; Stress; d-amphetamine
MeSH Terms: interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Second arm is placebo
  Interventions: Drug: Placebo
- 1 (Experimental): One arm is atomoxetine 40 mg per day
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 2
Drug: Atomoxetine — 20mg maximum of d-amphetamine
  Arms: 1

SUMMARY:
A total of 18 healthy volunteers will participate in this four-week, within-groups, double-blind, placebo-controlled study. The study has two phases separated by a 4 to 15-day washout period. Subjects will be randomly assigned to receive either 40 mg atomoxetine or placebo. For Phase I, subjects will be assigned to atomoxetine or placebo for 4 days. After receiving medication or placebo for three days, subjects will have a 6-hour laboratory session, where responses to physical and psychological stress of a 20 mg/70 kg (20 mg maximum) dose of d-amphetamine will be measured. Several physiological, hormonal, and subjective outcome measures will be obtained during the experimental sessions. Subjects will then have a 4-15 day washout period and will be crossed over to the alternative treatment for Phase II.

DETAILED DESCRIPTION:
Objective: This pilot study will examine the effects of a norepinephrine reuptake blocker, atomoxetine, on physiological and subjective responses to physical and psychological models of stress and oral amphetamine in healthy volunteers. The physical stress model will be the cold pressor test (CPT) and the psychological stress will be the paced auditory serial addition task (PASAT).

Our overall hypothesis is that atomoxetine treatment, compared to placebo, will attenuate the physiological and subjective responses to stress and d-amphetamine.

2. Research Design: Double-blind, placebo-controlled, within-groups, outpatient study.

3. Methodology: A total of 18 healthy volunteers will participate in this four-week, within-groups, double-blind, placebo-controlled study. The study has two phases separated by a 4 to 15-day washout period. Subjects will be randomly assigned to receive either 40 mg atomoxetine or placebo. For Phase I, subjects will be assigned to atomoxetine or placebo for 4 days. After receiving medication or placebo for three days, subjects will have a 6-hour laboratory session, where responses to physical and psychological stress of a 20 mg/70 kg (20 mg maximum) dose of d-amphetamine will be measured. Several physiological, hormonal, and subjective outcome measures will be obtained during the experimental sessions. Subjects will then have a 4-15 day washout period and will be crossed over to the alternative treatment for Phase II.

4. Findings: A total of 10 subjects have completed this study. This study has been published.

ELIGIBILITY:
Inclusion Criteria:

* Female and males, age 18 to 45 years
* Current history of good health and normal ECG
* For women: not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* History of heart disease, hypertension, renal or hepatic diseases, glaucoma, hyperthyroidism, or other medical conditions that the physician investigator deems as contraindicated for the patient to be in the study
* Current use of psychotropic medication(antidepressants, antipsychotics, or anxiolytics) and/or diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia and panic disorder within the past year.
* Current dependence on alcohol or on drugs or treatment for drug or alcohol addiction(amphetamines have greater abuse liability among those with drug addictions) within the past 5 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Measuring subjective responses to physical and psychological models of stress and oral amphetamine in healthy volunteers. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University